CLINICAL TRIAL: NCT05964101
Title: Neoadjuvant Anti-PD-1 Drug Nivolumab Combined With Chemotherapy in the Treatment of Primary Tracheal Squamous Cell Carcinoma
Brief Title: Nivolumab Combined With Chemotherapy in the Treatment of Primary Tracheal Squamous Cell Carcinoma
Acronym: GALAXY-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shuben Li, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2023-062-03
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Carcinoma, Squamous; Antineoplastic Agents
Keywords: tracheal tumor; neoadjuvant immunochemotherapy; surgery
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell; Tracheal Neoplasms | interventions — Nivolumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab (Experimental): Neoadjuvant treatment stage: Nivolumab 360mg, Carboplatin AUC5+ paclitaxel 100 mg/m ², iv, 3 weeks per cycle, 2-4 cycles in total; Surgical treatment stage: Patients with primary tracheal squamous cell carcinoma received radical surgery after neoadjuvant therapy, and patients who could not or refused surgical treatment due to various reasons were treated with multidisciplinary discussion.
  Interventions: Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: Nivolumab Injection [Opdivo] — Neoadjuvant treatment stage: Nivolumab +Carboplatin AUC+ paclitaxel
  Other Names: carboplatin; paclitaxel

SUMMARY:
This is a single-arm, open, II phase study to evaluate the safety and efficacy of Nivolumab + carboplatin + paclitaxel in 25 newly diagnosed patients with primary tracheal squamous cell carcinoma.

DETAILED DESCRIPTION:
Primary tracheal tumors are rare, comprising 0.01-0.4% of all cancer cases. Most airway tumors present with non-specific symptoms, such as shortness of breath and a sore throat, which may not be attributable to the tumors themselves, leading to diagnostic delay. With limited treatment options, surgical resection is considered the cornerstone therapy. Neoadjuvant therapy is recommended as standard treatment for the early stages (stage IB/II) and locally advanced stages (stage IIIA) of non-small cell lung cancer (NSCLC). Whether neoadjuvant therapy affects subsequent pathological or surgical outcomes of primary tracheal tumors remains unclear. This study aimed to characterize the outcomes of neoadjuvant therapy for the treatment of primary tracheal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Bronchoscopic biopsy confirmed as tracheal squamous cell carcinoma by pathological examination
2. PET-CT confirmed no metastasis;
3. ECOG physical status score 0-1;
4. Bronchoscopy, and chest CT is evaluated as early or locally advanced tracheal malignant tumor, and radical surgery is expected to be feasible or after neoadjuvant therapy.
5. Age ≥ 18 years;
6. Have one measurable lesion at least;
7. Good function of other major organs (liver, kidney, blood system, etc.):-absolute neutrophil count ((ANC) ≥ 1.5 × 109), platelet (≥ 100 × 109), hemoglobin (≥ 90g/L). Note: patients shall not receive blood transfusion or growth factor support within 14 days before blood collection during the screening period;-International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 × normal upper limit (ULN);-activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;- serum total bilirubin ≤ 1.5 × ULN (Gilbert syndrome patients with total bilirubin must be < 3×ULN). Fertile female patients with aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 × ULN, or liver metastasis with AST and ALT ≤ 5 × ULN
8. Fertile female patients must voluntarily take effective contraceptive measures more than 120 days after chemotherapy or the last administration of Nivolumab, whichever is later, and the urine or serum pregnancy test results less than 7 days before entering the group were negative. Unsterilized male patients must voluntarily take effective contraceptive measures ≥ 120 days after chemotherapy or the last administration of Nivolumab, whichever is the latter.
9. Sign informed consent;

Exclusion Criteria:

1. Any Chinese herbal medicine used to control cancer was used within 14 days before the first administration of the study drug;
2. Patients with other malignant tumors in the five years before the start of this trial.
3. Complicated with unstable systemic diseases, including active infections, uncontrolled hypertension, unstable angina pectoris, congestive heart failure [higher than II (New York College of Cardiology)], severe arrhythmias, liver, kidney or metabolic diseases;
4. Active, known or suspected autoimmune diseases, or autoimmune paraneoplastic syndrome requiring systemic treatment;
5. A history of active bleeding or embolism within 6 months, or received thrombolysis or anticoagulation therapy, or the researchers believe that there is an obvious tendency of gastrointestinal bleeding (such as esophageal varices have the risk of bleeding, local active ulcer lesions, etc.);
6. Had is suffering from nephrotic syndrome
7. Allergic to experimental drugs;
8. Complicated with HIV infection or active hepatitis.
9. Vaccination within 4 weeks before the start of this trial;
10. Those who had undergone other major operations or severe injuries within the previous 2 months;
11. Clinically uncontrolled pleural effusion or ascites requiring pleural or abdominal puncture drainage within 2 weeks before admission;
12. Pregnant or lactating women;
13. Those with neurological diseases or mental disorders.
14. Participated in another therapeutic clinical study at the same time;
15. Other researchers did not consider it appropriate to enroll in the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | up to 4 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery
Safety: frequency of severe adverse events | up to 5 months
  The frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  PFS is defined as the time from the enrollment of the subject to the first determination of disease progression or death of any cause according to RECISTv1.1, whichever occurs first.
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Disease control rate (DCR) | up to 60 months
  The proportion of patients whose best overall remission (BOR) is CR, PR or disease stable (SD) according to RECISTv1.1 evaluation
Duration of remission (DOR) | up to 60 months
  According to the time from the first recording of objective remission to relapse or death from any cause determined by RECISTv1.1, whichever occurs first.
R0 rate | up to 4 months
  There were no visible tumors in the surgical margin, and the tumor cells in the surgical margin within 1mm were negative under the microscope

CONTACTS AND LOCATIONS:
Overall Officials: Shuben Li, PhD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided